CLINICAL TRIAL: NCT03554577
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2018_12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_12
Record Dates: First submitted 2018-05-07; First posted 2018-06-13 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with each sound changing principle (Noise Reduction principle (NR)) in a randomized order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hearing Aid without NR (Active Comparator): Hearing Aid without Noise Reduction (NR) serves as reference condition.
  Interventions: Device: Hearing Aid without NR
- Hearing Aid with NR_A (Experimental): NR_A: Noise Reduction principle A
  Interventions: Device: Hearing Aid with NR_A
- Hearing Aid with NR_B (Experimental): NR_B: Noise Reduction principle B.
  Interventions: Device: Hearing Aid with NR_B
- Hearing Aid with NR_C (Experimental): NR_C: Noise Reduction principle C.
  Interventions: Device: Hearing Aid with NR_C

INTERVENTIONS:
Device: Hearing Aid without NR — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs.
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Other Names: NR: Noise Reduction
  Arms: Hearing Aid without NR
Device: Hearing Aid with NR_A — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs.
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Other Names: NR_A: Noise Reduction principle A
  Arms: Hearing Aid with NR_A
Device: Hearing Aid with NR_B — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs.
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Other Names: NR_B: Noise Reduction principle B
  Arms: Hearing Aid with NR_B
Device: Hearing Aid with NR_C — Each participant will be fitted with the 4 different Noise Reduction (Sound Changing) principles on the same hearing aid, saved to 4 manual programs.
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Other Names: NR_C: Noise Reduction principle C
  Arms: Hearing Aid with NR_C

SUMMARY:
A methodical evaluation of novel sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and asses strength and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Both, objective laboratory measurements as well as subjective evaluations in real life environment will be carried out. This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders
* colour blinded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Sound quality ratings | 4 weeks
  The sound quality ratings will be assessed with the aid of a Multi-Stimulus Test. The data, serving as the primary outcome measure, are collected in the laboratory and will use a continuous rating scale. The scale ranges from 0 "very bad" to 100 "very good" in increments of 1.

SECONDARY OUTCOMES:
Oldenburg sentence test in noise | 4 weeks
  The data, serving as secondary outcome is a Signal to noise ratio (SNR) in decibel (dB) where a 50% speech reception threshold is reached. This outcome measurement will be carried out in the laboratory.
Oldenburg sentence test & manual tracking task | 4 weeks
  A dual task paradigm will be used in which the Oldenburg Sentence test in noise will be administered as a primary task, and the subject will manually track a point on a computerised elliptical track as a secondary task. The aim is to recall as many words from the presented sentence at a predefined SNR and track the point as accurately as possible at the same time. The SNR is set as the level at which a subject reaches a speech reception threshold of 80-90%. The data derived, serving as a secondary outcome measure, are a [%] of time on target and distance error from the target.
Adaptive Categorial Listening Effort Scaling (ACALES) | 2 weeks
  The ACALES procedure determines self-reported individual listening effort on a scale from "extreme effort" to "no effort" within a signal-to-noise ratio range that corresponds to individual subject perceptions.
  The data, serving as a secondary outcome, are a set of points on a categorial scale (subjectively perceived listening effort) as a function of different SNRs.
Self-report form | One week
  A qualitative questionnaire with predefined questions and comment sections to gather information on individual perceptions regarding the comparison of two different hearing programs during different laboratory-based acoustic scenes. For details of the hearing aid settings, see study arms. The data collected from this questionnaire are scores on a continuous rating scale ranging from "hearing program A is much worse than hearing program B" to "hearing program B is much better than hearing program A" and any subjective comments given.

OTHER OUTCOMES:
Interaural Phase Difference (IPD) Detection thresholds | 1 week
  A 2 Interval - 2 Alternative Forced Choice task to measure the psychometric function of IPD detection with changing stimulus frequency. The data, serving as an outcome measure, is the individual interaural phase difference (IPD) frequency threshold (the frequency up to which 75% correct answers are given).
Non-verbal Trail Making Test A & B | 1 week
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The data, serving as an outcome measure, are time-to-complete the set in seconds.
color-word-interference test by J.R.Stroop | 1 week
  The color-word- interference test ("Farb-Wort-Interferenztest nach J.R.Stroop" (version: "Günther Bäumler")) is a neuropsychological test of visual attention and interferer suppression and will be carried out in the laboratory. In the first trial, the subject has to read the names of colours written on a card as fast and accurately as possible. In the second trial, the subject has to name the colour ink of filled boxes on a card as quickly and accurately as possible. In the third trial, the names of colours are written on a card in a dissimilarly coloured ink. The participant must read aloud the written words, whilst ignoring the colour of the ink. The data, serving as an outcome measure, are time-to-complete the sets in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Raether, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No